CLINICAL TRIAL: NCT05441865
Title: The Influence and Potential Mechanism of Cardiovascular Risk Factors on the Cognitive Trajectories Among Cognitively Intact Older Adults
Brief Title: Cardiovascular Risk Factors and Cognitive Trajectories
Status: Completed | Type: Observational
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Xiaozhen LV, Associate Researcher, Peking University Sixth Hospital
Other Study IDs: 82003539
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-04

CONDITIONS: Normal Cognition; Cardiovascular Risk Factors; Cognitive Change; Cerebral Blood Flow; FMRI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cognitive trajectory cohort: Th cognitive trajectory cohort, based on CLHLS dataset, will be used to evaluate the influence of cardiovascular risk factors on the cognitive trajectories among cognitively intact older adults
- neuroiming sample: The neuroiming sample, including cognitively intact older adults with MRI data, will be used to explore the potential mechanism of the cardiovascular risk factors and cognitive function.

SUMMARY:
The cognitive trajectory varies among non-demented older adults. In a 12-year follow-up study, we found approximately 5% participants presented rapid cognitive decline. Cardiovascular diseases increased the risk of cognitive decline. However, the influence of cardiovascular risk factors on cognitive decline remained inconsistent. Besides, the potential mechanism of the cardiovascular risk factors and cognitive function has not been fully investigated. Therefore, the proposed program will include two sub-studies. The first sub-study will use the longitudinal data from the Chinese Longitudinal Healthy Longevity Survey to evaluate the influence of cardiovascular risk factors on the trajectories of cognitive function. The second sub-study will recruit cognitive intact older adults with different levels of cardiovascular risk factors. The association among cardiovascular risk factors, cerebral blood flow, brain functional connectivity and cognitive function will be investigated with structural equation modeling. The findings of the proposed program will provide novel insight on preventing cognitive decline from the angle of maintaining healthy vascular function, and will provide evidence in elucidating the potential neurovascular mechanism between cardiovascular risk factors and cognitive function.

ELIGIBILITY:
For the cognitive trajectory cohort (the data had been collected):

Inclusion Criteria:

1. Aged 65 or over at baseline;
2. With normal cognitive function at baseline (score ≥ 18 on the Chinese version of Mini-Mental State Examination, MMSE);
3. Had at least one domain information about cardiovascular risk factors (hypertension, diabetes, dyslipidemia, obesity, exercise, diet and smoking) at baseline;
4. Completed cognitive function assessment at least twice during 3 waves following-up after baseline;
5. Provided informed consent voluntarily.

Exclusion Criteria:

1. Aged <65;
2. had a history of dementia or MMSE score < 18 at baseline;
3. Without more than once cognitive function assessment during the follow-up;
4. Refused to participate the survey.

For the neuroimaging sample, who would be enrolled by this study:

Inclusion Criteria:

1. Aged 55-80;
2. Right-handed;
3. Primary school education or above, with normal communication ability;
4. No complaints of cognitive impairment or decline;
5. MMSE score ≥ 26;
6. Clinical dementia rating (CDR) =0;
7. Provided informed consent voluntarily.

Exclusion Criteria:

1. Severe visual or hearing impairment, difficult to complete cognitive function assessment;
2. Had contraindications to magnetic resonance examination, such as claustrophobia, cardiac pacemaker and artificial heart valve;
3. Had cardiovascular diseases (such as myocardial infarction and unstable angina pectoris), severe respiratory diseases, malignant tumors, renal failure and other serious physical diseases;
4. Had diseases that could affect cognitive function, such as hypothyroidism, syphilis, vitamin B12 deficiency and anemia;
5. Had a history of any mental disease;
6. Had a history of cerebrovascular disease, or obvious space occupying lesions in the brain revealed by magnetic resonance examination;
7. Refused to participate the survey.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the cognitive trajectory cohort, the study population was those community-dwelling older adults with normal cognitive function, completed at least one domain information about cardiovascular risk factors at baseline, and completed cognitive function assessment at least twice during 3 waves following-up after baseline.
  For the neuroimaging sample, the study population was those community-dwelling older adults with normal cognitive function, without severe physical disease and mental disorders, could complete cognitive function assessment and MRI examination.
Sampling Method: Non-Probability Sample
Enrollment: 3372 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Regression coefficients | up to 10 years
  the influence of cardiovascular risk factors on cognitive change

SECONDARY OUTCOMES:
the correlation coefficient | baseline
  the relationship among cognitive function score, value of cerebral blood flow, and functional connectivity strength

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhen Lv, Principal Investigator — Peking University Six Hospital
Locations (1):
- Peking University Six Hospital, Beijing, China